CLINICAL TRIAL: NCT02782039
Title: Register of Patients With Anti-Phospholipids Syndrome (APS) and/or Systemic Lupus Erythematosus (SLE)
Acronym: SAPL-LUPUS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI15010
Record Dates: First submitted 2015-11-11; First posted 2016-05-25 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Anti-Phospholipids Syndrome (APS); Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Antiphospholipid Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of that register is to collect medical information about patients suffering of APS with or without associated SLE.

DETAILED DESCRIPTION:
Recruitment of patients with APS and SLE treated. Retrospective and prospective register.

ELIGIBILITY:
Inclusion Criteria:

* Patient with APS
* Patient with SLE

Exclusion Criteria:

* Dependent person
* Hospitalized without consent and not protected by law
* Detainee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering of APS with or without associated SLE
Sampling Method: Non-Probability Sample
Enrollment: 868 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients enrolled with Anti-Phospholipids syndrome (APS) and/or Systemic Lupus Erythematosus (SLE) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Costedoat-Chalumeau, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Cochin, Paris, PARIS
  - Hôpital Claude Huriez, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariette F, Le Guern V, Nguyen Y, Yelnik C, Morel N, Hachulla E, Lambert M, Guettrot-Imbert G, Mouthon L, Ebbo M, Costedoat-Chalumeau N. Cluster analysis of clinical manifestations assigns systemic lupus erythematosus-phenotype subgroups: A multicentre study on 440 patients. Joint Bone Spine. 2024 Dec;91(6):105760. doi: 10.1016/j.jbspin.2024.105760. Epub 2024 Jul 6. PMID 38972539
- [Derived] Dupre A, Morel N, Yelnik C, Moguelet P, Le Guern V, Stammler R, Nguyen Y, Paule R, Dufrost V, Ackermann F, Benhamou Y, Godeau B, Lambert M, Duffau P, Mekinian A, Saadoun D, Mouthon L, Hachulla E, Maillard H, Levesque H, Morell-Dubois S, Leroux G, Piette JC, Chasset F, Costedoat-Chalumeau N. Cutaneous Involvement in Catastrophic Antiphospholipid Syndrome in a Multicenter Cohort of 65 Patients. JAMA Dermatol. 2023 Jan 1;159(1):62-67. doi: 10.1001/jamadermatol.2022.5221. PMID 36477813
- [Derived] Morel N, Bonnet C, Mehawej H, Le Guern V, Perard L, Roumier M, Brezin A, Godeau B, Haroche J, Benhamou Y, Lambert M, Yelnik CM, Maillard N, Bodaghi B, Piette JC, Costedoat-Chalumeau N. CATASTROPHIC ANTIPHOSPHOLIPID SYNDROME AND POSTERIOR OCULAR INVOLVEMENT: Case Series of 11 Patients and Literature Review. Retina. 2021 Nov 1;41(11):2332-2341. doi: 10.1097/IAE.0000000000003185. PMID 33840791